CLINICAL TRIAL: NCT03100591
Title: Single-center, Open-label Study With 14C-radiolabeled ACT-132577 to Investigate the Mass Balance, Pharmacokinetics, and Metabolism Following Single Oral Administration to Healthy Male Subjects
Brief Title: A Study to Evaluate ACT-132577 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC-080-104
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — aprocitentan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 14C-radiolabelled ACT-132577 (Experimental): On Day 1, subjects will receive a single oral dose of 25 mg 14C-radiolabeled ACT-132577, administered as an oral formulation in the fasted state
  Interventions: Drug: 14C-radiolabeled ACT-132577

INTERVENTIONS:
Drug: 14C-radiolabeled ACT-132577 — Single oral dose of 3.7 megabecquerel (MBq) (100 microcurie [μCi]) 14C-radiolabeled ACT-132577 administered as 1 capsule of 25 mg
  Other Names: Aprocitentan

SUMMARY:
The primary purpose of this study is to investigate the rate and routes (urine and feces) of elimination of ACT-132577, and the mass balance in urine and feces

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure;
* Healthy male subjects aged between 45 and 65 years (inclusive) at screening;
* Body mass index of 18.0 to 28.0 kg/m2 (inclusive) at screening;
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests.

Exclusion Criteria:

* Values of hepatic aminotransferase (alanine aminotransferase and/or aspartate aminotransferase) > 3 × upper limit of normal range at screening;
* Hemoglobin < 100 g/L at screening;
* Known hypersensitivity to ACT-132577 or drugs of the same class, or any excipient of the ACT-132577 drug formulation;
* Known hypersensitivity or allergy to natural rubber latex;
* Previous exposure to ACT-132577;
* Treatment with another investigational drug within 3 months prior to screening or participation in more than 4 investigational drug studies within 1 year prior to screening;
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol;
* A radiation burden of > 0.1 milliSievert (mSv) and ≤ 1.0 mSv in the period of 1 year prior to screening; a radiation burden of ≥ 1.1 mSv and ≤ 2.0 mSv in the period of 2 years prior to screening, etc. (add 1 year per 1 mSv).

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion of radioactivity in urine and feces | From study treatment administration up to day 15
  14C-radioactivity will be measured daily in urine and feces samples for determination of total radioactivity recovery

SECONDARY OUTCOMES:
Number of subjects with treatment-emergent adverse events and serious adverse events | From study treatment administration up to day 32
  Collection of any adverse event at each dose level
Maximum plasma concentration (Cmax) of 14C-radiolabeled ACT-132577 | From study treatment administration up to day 15
  Cmax is directly derived from the observed plasma concentrations of ACT-132577 and its metabolites
Time to reach Cmax (tmax) of 14C-radiolabeled ACT-132577 | From study treatment administration up to day 15
  tmax is directly derived from the observed plasma concentrations of ACT-132577 and its metabolites
Terminal half-life (t1/2) of 14C-radiolabeled ACT-132577 | From study treatment administration up to day 15
  t1/2 is calculated from the terminal rate constant obtained from the plasma concentrations-time curves of ACT-132577 and its metabolites
Area under the plasma concentration-time curve (AUC) of 14C-radiolabeled ACT-132577 | From study treatment administration up to day 15
  AUC is defined for the time intervals from zero to time t of the last measured concentration above the limit of quantification and from zero to infinity
Maximum plasma concentration (Cmax) of ACT-132577 and its metabolites | From study treatment administration up to day 15
  Cmax is directly derived from the observed plasma concentrations of ACT-132577 and its metabolites
Time to reach Cmax (tmax) of ACT-132577 and its metabolites | From study treatment administration up to day 15
  tmax is directly derived from the observed plasma concentrations of ACT-132577 and its metabolites
Terminal half-life (t1/2) of ACT-132577 and its metabolites | From study treatment administration up to day 15
  t1/2 is calculated from the terminal rate constant obtained from the plasma concentrations-time curves of ACT-132577 and its metabolites
Area under the plasma concentration-time curve (AUC) ACT-132577 and its metabolites | From study treatment administration up to day 15
  AUC is defined for the time intervals from zero to time t of the last measured concentration above the limit of quantification and from zero to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- PRA Health Sciences, Groningen, Netherlands